CLINICAL TRIAL: NCT04877951
Title: Postural Control in Stance and During Functional Mobility Following Management of Parkinson's Disease With LSVT BIG Training
Brief Title: PC in Stance and During Functional Mobility Following BIG for PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Patti Berg-Poppe, Associate Professor, University of South Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC in PD after BIG
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
Keywords: postural control; gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Effect of LSVT BIG therapy on Postural Control and Gait Parameters (Other): LSVT BIG is a commonly used protocol to manage functional movement for those with Parkinson's Disease. This study measured postural control and gait parameters following a 4-week course of LSVT BIG therapy.
  Interventions: Behavioral: LSVT BIG

INTERVENTIONS:
Behavioral: LSVT BIG — LSVT BIG is a 4-week program that focuses on movement recalibration for people with a diagnosis of Parkinson's disease.

SUMMARY:
LSVT BIG is an intensive, amplitude based rehabilitation program that has been demonstrated to improve one of the hallmark features of Parkinson's disease, specifically bradykinesia. We are interested in knowing the effects of this therapeutic approach on postural control and gait parameters.

DETAILED DESCRIPTION:
LSVT BIG is an intensive, amplitude based rehabilitation program that has been demonstrated to improve one of the hallmark features of Parkinson's disease, specifically bradykinesia. Postural instability and gait disturbance is another debilitating feature of Parkinson's disease. While LSVT BIG targets postural correction through exercises which challenge balance, the effect of this intervention on stability margins and functional balance assessments have not been well established in the literature. This study includes outcome measures not previously examined with this intervention and may provide valuable evidence regarding the impact of this intervention on postural control, balance and falls risk. Alternative amplitude programs have also been designed to meet the needs of patients with PD. These programs adjust frequencies for patients and individualize sessions more than LSVT BIG. We are interested in knowing if these alternative frequencies and amplitude approaches are similarly as effective as LSVT BIG in our outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included in the study if they have been diagnosed with idiopathic Parkinson's disease and are English speaking.

Exclusion Criteria:

* Exclusion Criteria: 1) previous completion of LSVT BIG or other formal amplitude program training 2) non-idopathic Parkinsonism 3) any medical condition that would contraindicate exercise (ie. unstable cardiovascular disease) 4) cognitive impairment that limits ability to follow direction or demonstration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mini Balance Evaluation Systems Test (Mini-BESTest) | Pre-Intervention (baseline) and Post-Intervention (week 5)
  A change in reactive, proactive, and sensory contributions to postural control (balance) is assessed.
Fullerton Advanced Balance Scale (FAB) | Pre-Intervention (baseline) and Post-Intervention (week 5)
  A change in higher level assessment of postural control is assessed.
Functional and Multidirectional Reach Tests | Pre-Intervention (baseline) and Post-Intervention (week 5)
  A change in proactive postural control strategies is assessed.
Center of Pressure measures (digitized walkway) | Pre-Intervention (baseline) and Post-Intervention (week 5)
  A change in the limits of stability is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Patti J Berg-Poppe, PhD, Principal Investigator — University of South Dakota